CLINICAL TRIAL: NCT07274033
Title: Effect of Manual Lymphatic Drainage on Muscle Fatigue in Female 11-a-side Football Players
Acronym: EDLMF11
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Principal Investigator, Edurne Úbeda D'Ocasar, Doctor Edurne Úbeda D'Ocasar, Camilo Jose Cela University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UCJCDLMF
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Women
Keywords: Manual Lymphatic Drainage; Football; Women

STUDY DESIGN:
Masking Description: One of the members of the research team that will carry out the data analysis is not aware of the intervention that will be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual Lymphatic Drainage Group (Experimental): The study consists of three visits. During the first visit, participants are informed about the study, eligibility criteria are verified, informed consent is obtained, and baseline assessments are conducted using psychophysiological questionnaires and thigh circumference measurements. In the second visit, assessments are repeated and fatigue is induced through guided squats at 50-60% of estimated 1RM, monitored via a linear encoder. Fatigue is defined as a 20% loss in execution velocity. Immediately after fatigue induction, manual lymphatic drainage (MLD) is applied for 10 minutes (5 minutes per quadriceps), following Emil Vodder's standardized technique. Post-intervention, performance testing and measurements are repeated. The third visit, conducted 15 days later, serves as a follow-up to evaluate sustained effects without further intervention, repeating the fatigue protocol and all assessments.
  Interventions: Other: Manual lymphatic draige

INTERVENTIONS:
Other: Manual lymphatic draige — This method, part of complex decongestive physiotherapy, involves gentle massage techniques that stimulate lymphatic circulation and venous return. MLD promotes lymph fluid mobilization, increases lymphangiomotor activity, and has positive effects on the immune system. Its application has shown to reduce limb edema, decrease muscle fatigue, and raise pain thresholds. Moreover, the gentle touch during MLD activates cutaneous receptors that influence the parasympathetic nervous system, producing physiological changes such as reduced heart rate, blood pressure modulation, and increased muscle strength.

SUMMARY:
This clinical trial investigates the effectiveness of manual lymphatic drainage (MLD) in accelerating recovery following induced fatigue in female football players. The study integrates objective performance measurements using linear encoders with anthropometric assessments and psychophysiological evaluations. It aims to quantify the impact of MLD on neuromuscular recovery, muscle edema, and perceived fatigue, considering sex-specific physiological factors and the influence of sleep and psychological stress. The findings will contribute to developing non-invasive, individualized recovery strategies to enhance performance and reduce injury risk in women's football.

DETAILED DESCRIPTION:
This study aims to assess the effectiveness of manual lymphatic drainage (MLD) as a recovery strategy following induced fatigue in female football players. The intervention is applied immediately after a standardized fatigue protocol using a linear encoder to objectively measure performance decline. The study adopts a multidimensional approach, integrating biomechanical, physiological, and psychometric variables to evaluate recovery.

Participants will undergo three experimental sessions involving a fatigue protocol followed by either MLD or control conditions. Performance will be assessed through guided machine squats, measuring the number of repetitions and time until a 20% velocity loss. Thigh circumference will be measured pre- and post-intervention to monitor fluid shifts and potential edema. Subjective recovery perception will be recorded, and emotional state will be evaluated using the Hospital Anxiety and Depression Scale (HADS). Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) to explore its influence on fatigue and recovery response.

This trial addresses the need for non-invasive, efficient recovery strategies tailored to female athletes, considering sex-specific physiological and psychological factors. The findings may contribute to optimizing post-exercise recovery protocols and reducing injury risk in women's football.

ELIGIBILITY:
Inclusion Criteria:

* Female athletes actively participating in 11-a-side football, either federated or official team members.
* Age ≥ 16 years to 20 years old.
* Regular training (≥ 3 sessions per week) or active competition
* No food intake within 3 hours prior to evaluation (to standardize the influence of digestion on performance).
* No acute lower limb injury in the past 3 months.
* Availability to attend all three study visits.
* Signed informed consent; for participants under 18, parental consent is also required.

Exclusion Criteria:

* History of deep vein thrombosis
* Decompensated heart failure
* Active lower limb infection
* Pregnancy
* Recent lower limb surgery (< 3 months), or any medical contraindication to receiving manual lymphatic drainage (MLD).
* Failure to comply with the fasting requirement prior to performance testing.

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of repetitions | baseline; 5 minutes before and 5 minutes after the first procedure, 5 minutes before and 5 minutes after the second procedure, and 15 days after the procedure was completed.
  Number of repetitions until 20% velocity loss: recorded via linear encoder during guided squat test.
Time to fatigue | baseline; 5 minutes before and 5 minutes after the first procedure, 5 minutes before and 5 minutes after the second procedure, and 15 days after the procedure was completed.
  Time to fatigue (seconds): total time from first repetition until velocity drops by 20%.
Velocity profile | baseline; 5 minutes before and 5 minutes after the first procedure, 5 minutes before and 5 minutes after the second procedure, and 15 days after the procedure was completed.
  average velocity per repetition, expressed in m/s.
Thigh circumference (cm) | baseline; 5 minutes before and 5 minutes after the first procedure, 5 minutes before and 5 minutes after the second procedure, and 15 days after the procedure was completed.
  measured with a non-elastic tape at the midpoint between the anterior superior iliac spine and the upper border of the patella, in both legs, pre- and post-intervention.
Perceived fatigue | baseline; 5 minutes before and 5 moinutes after the first procedure, 5 minutes before and 5 minutes after the second procedure, and 15 days after the procedure was completed.
  assessed using Borg CR-10 scale (0 = no fatigue, 10 = maximum fatigue).
Perceived pain (VAS) | baseline; 5 minutes before and 5 minutes after the first procedure, 5 minutes before and 5 minutes after the second procedure, and 15 days after the procedure was completed.
  assessed using Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (maximum pain).
Perceived recovery (PRS) | baseline; 5 minutes before and 5 minutes after the first procedure, 5 minutes before and 5 minutes after the second procedure, and 15 days after the procedure was completed.
  assessed using the Perceived Recovery Status Scale (PRS), ranging from 0 (no recovery) to 10 (full recovery).

SECONDARY OUTCOMES:
Sleep quality (PSQI) | baseline, after the second procedure and 15 days after the procedure was completed
  assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item questionnaire with scores ranging from 0 to 21 (higher scores indicate poorer sleep quality).
Emotional state | baseline, after the second procedure and 15 days after the procedure was completed
  assessed using the Hospital Anxiety and Depression Scale (HADS), comprising 14 items across anxiety and depression subscales (scores range from 0 to 21 per subscale).
Sociodemographic Variables | Baseline
  Age, Height, Body weight, Body mass Index
Dominant leg | Baseline
  self-reported (leg used to kick the ball).
Sports experience (years) | baseline
  total years of systematic football practice.
Training frequency (sessions/week) | baseline
  average number of sessions during the season.
Menstrual cycle phase | baseline, after the second procedure and 15 days after the procedure was completed
  self-reported, to control for physiological variations in fatigue and recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Úbeda Docasar, Doctor, Principal Investigator — University Camilo José Cela
Locations (1):
- University of Camilo José Cela, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
What IPD Will Be Shared:
  De-identified individual participant data (IPD) related to primary and secondary outcome measures, including performance metrics (e.g., number of repetitions, velocity profiles), anthropometric data (e.g., thigh circumference), and questionnaire responses (e.g., Borg scale, VAS, PRS, PSQI, HADS).
  When Will IPD Be Available:
  IPD will be made available upon publication of the main results or within 12 months after study completion.
  How Will IPD Be Shared:
  Data will be shared upon reasonable request to the principal investigator. Access will be granted for academic and non-commercial research purposes, following approval by the ethics committee and under a data-sharing agreement to ensure confidentiality and compliance with GDPR.
  With Whom:
  Qualified researchers affiliated with academic institutions or research organizations.